CLINICAL TRIAL: NCT04660786
Title: Intralesional Vitamin D3 Injection in Treatment of Alopecia Areata: A Novel Approach
Brief Title: Intralesional Vitamin D in Alopecia Areata
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Alexandria University (Other)
Responsible Party: Principal Investigator, marwa eldeeb, lecturer of dermatology, Alexandria University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 0304857
Record Dates: First submitted 2020-12-03; First posted 2020-12-09 (Actual); Last update posted 2021-07-26 (Actual); Status verified 2021-07

CONDITIONS: Alopecia Areata
MeSH Terms: conditions — Alopecia Areata | interventions — Triamcinolone Acetonide; Vitamin D

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- intralesional injection of triamcinolone acetonide (Active Comparator): 5mg/ml) using sterile saline for dilution every 4 weeks for 3 sessions
  Interventions: Drug: triamcinolone acetonide
- intralesional injection of vitamin D (Active Comparator): (2.5 mg/mL) every 4 weeks for 3 sessions
  Interventions: Drug: vitamin D

INTERVENTIONS:
Drug: triamcinolone acetonide — local immunosuprresent
  Arms: intralesional injection of triamcinolone acetonide
Drug: vitamin D — local immunomodulator
  Arms: intralesional injection of vitamin D

SUMMARY:
To evaluate the efficacy and safety of intralesional injection of vitamin D3 versus intralesional injection of corticosteroids in treatment of alopecia areata.

this will be carried out on 40 patients who attend hair outpatient clinic, department of dermatology, Faculty of medicine, Alexandria University, Egypt.

The patients will be randomly assigned into two groups (A and B), each group contains 20 patients. Patients will be blindly subjected to intralesional injection of triamcinolone acetonide (5mg/ml) using sterile saline for dilution every 4 weeks for 3 sessions (11,12) or intralesional injection of vitamin D (an aqueous preparation of cholecalciferol (Devarol® ampoule 200,000 IU/2 mL, Memphis, Egypt) (2.5 mg/mL) every 4 weeks for 3 sessions. The maximum total amount of vitamin D3 injected into a patient in 1 session will be 5 mg Injection will be preceded by topical anaesthesia under occlusion for 30 minutes.

ELIGIBILITY:
Inclusion Criteria:

Site: scalp. Extent: localized alopecia areata (less than 50% scalp involvement).

Exclusion Criteria:

1. Other skin diseases affecting the scalp
2. Pregnant or lactating women.
3. Bleeding or coagulation disorders
4. Immunocompromised patients.
5. Known hypersensitivity to vitamin D3.
6. Patients who received systemic or topical treatment for alopecia areata in the last month.
7. Patients taking vitamin D supplements in the last 6 months.
8. Patients treated with topical vitamin D analogues.
9. Patients with diseases known to alter vitamin D level as autoimmune diseases, liver or renal diseases.
10. Obesity (defined as body mass index ≥ 25).

Min Age: 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2021-11-01 (Estimated); Primary Completion 2022-12-01 (Estimated); Study Completion 2022-12-01 (Estimated)

PRIMARY OUTCOMES:
Regrowth Score (RGS) | three month
  calculation at week 12 using a 5-point semiquantitative score (RGS)(0 = regrowth < 10%; 1 = regrowth 11- 25%; 2 = regrowth26 - 50%; 3 = regrowth 51- 75%; 4: regrowth > 75%)

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Medicine, Alexandria, Egypt

IPD SHARING:
Plan to Share IPD: No